CLINICAL TRIAL: NCT02302014
Title: Randomised Trial of Early Versus Delayed Future Care Planning for Patients and Families Living With Advanced Heart Disease
Brief Title: Palliative Care for Patients With Advanced Heart Disease
Acronym: FLAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Marie Curie FLAME trial
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Acute Coronary Syndrome; Congestive Cardiac Failure; Palliative Care
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palliative Care Intervention (Experimental): Baseline interview with trial cardiologist and trial nurse lasting for up to 1 hour Creation of a Future Care Plan (FCP) document following this baseline interview Sharing of FCP document with primary care and unscheduled care organisations 6 week interview with trial nurse lasting for up to 1 hour to review FCP 12 week interview with trial nurse lasting for up to 1 hour to review FCP Continuous access to trial nurse by mobile telephone 9am - 5pm Monday-Friday for 12 weeks Trial nurse will - ensure FCP is appropriately shared with primary and secondary care, patient is registered on primary care palliative care register and will liaise with specialist PC services and the general practitioner as needed.
  Interventions: Other: Palliative Care Intervention
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Other: Palliative Care Intervention — Baseline interview with trial cardiologist and trial nurse lasting for up to 1 hour Creation of a Future Care Plan (FCP) document following this baseline interview Sharing of FCP document with primary care and unscheduled care organisations 6 week interview with trial nurse lasting for up to 1 hour to review FCP 12 week interview with trial nurse lasting for up to 1 hour to review FCP Continuous access to trial nurse by mobile telephone 9am - 5pm Monday-Friday for 12 weeks Trial nurse will - ensure FCP is appropriately shared with primary and secondary care, patient is registered on primary care palliative care register and will liaise with specialist PC services and the general practitioner as needed.
  Arms: Palliative Care Intervention

SUMMARY:
Patients admitted as an unscheduled hospital admission with either a acute heart failure syndrome (ACF) or acute coronary syndrome (ACS) will be eligible if their 6-12 month mortality risk is estimated to be 20% or greater at the time of discharge. Mortality risk is estimated using GRACE (for ACS) or EFFECT (for AHF) scores. Patients are randomly allocated to receive a holistic care intervention based around the creation of a detailed Future (anticipatory) Care Plan which is agreed with the patient and their family and which is shared with the Family Doctor and Emergency Services including ambulance teams. Primary endpoint is quality of life assessed by questionnaire.

DETAILED DESCRIPTION:
Patients with either acute coronary syndrome(ACS) or acute heart failure (AHF) achieving an estimated risk of mortality within 12 months of 20% or greater (GRACE score for ACS and EFFECT score for AHF) will be assigned to early or delayed intervention using a web-based randomisation system.

Inclusion criteria:

Age > 18 years Unscheduled hospital admission due to congestive heart failure and or acute coronary syndrome 12 month estimated mortality risk of 20% or greater Optimal tolerated medical and device therapy

Exclusion criteria:

Expected survival < 28 days Other life limiting non-cardiac condition likely to cause death within 12 months Moderate or severe dementia Moderate or severe cognitive impairment

Supportive & Palliative Care Planning Intervention The planned intervention will follow the core principles of holistic palliative care. The detailed content may be adapted following the baseline qualitative interviews and focus group study outlined above and may evolve during the pilot phase (see below).

The first component of the intervention will consist of an interview with the patient and carer within 7 days of enrolment This will be undertaken by the trial consultant cardiologist and the trial nurse in a quiet room either in the hospital or in the patients home. This baseline consultation will explore the clinical and social needs of the patient and their carer, previous and current clinical status and treatment, goals of treatment and care now and in event of a future clinical deterioration, and cardiopulmonary resuscitation (CPR) status. The aim will be to develop a patient-centred Future Care Plan (FCP). This interview will also establish whether the patient and carer are happy to share the FCP with the community-based care team and out-of-hours emergency care services.

Two further scheduled patient/carer consultations with the nurse specialist will take place at 6 and 12 weeks following enrolment and will explore issues around cardiac care, physical, social, psychological, spiritual, cultural and information needs. At each of these meetings the FCP will be reviewed in detail and any changes will be made to a new document which will be shared with other organisations as outlined above with the patient's permission.

The second component of the intervention is continuous supportive care delivered by the trial nurse specialist who will act as professional carer and advocate for the patient during the 12 week intervention phase. Specifically, the nurse will be available on a mobile phone Monday to Friday, 0900 to 1700 for the patient or carer to call for advice or support. This trial nurse will ensure that the patient is placed on the primary care palliative care register. They will also provide opportunities for the patient and their family to ask for information about their condition and care, and that their current FCP is available to primary care, out-of-hours services and on the hospital patient information systems and updated at no less than 6 weekly intervals. The nurse will review the details of the FCP with the patient at each follow-up interview focusing on changes in the patient's symptoms, treatment goals, cardiopulmonary resuscitation status and preferences for place of care should they deteriorate.

The trial nurse will work closely with the palliative care team, the trial cardiologist and the patient's general practitioner. In order to document the success of this interface process, the nurse will document the number, duration and content of each communication with these healthcare professionals as they arise during the study.

The trial nurse specialist will use an established tool to monitor and document patient and carer needs at each visit using a Needs Assessment Tool for Palliative Care. The patient's secondary and primary care teams will be informed of the patient's involvement in the trial. Since some patients may choose not to take-up the services defined within the intervention we will carefully document their utilisation of the interventional services offered. Use of primary care services will be carefully monitored during the study period. All clinical data including comorbidities will be documented at the time of enrolment in the study.

Summary of the intervention: patients will be randomised while in hospital to either early intervention for 12 weeks or delayed intervention which will start 12 weeks after discharge, this too will last for 12 weeks.

INTERVENTION

Baseline interview with trial cardiologist and trial nurse lasting for up to 1 hour Creation of a Future Care Plan (FCP) document following this baseline interview Sharing of FCP document with primary care and unscheduled care organisations 6 week interview with trial nurse lasting for up to 1 hour to review FCP 12 week interview with trial nurse lasting for up to 1 hour to review FCP Continuous access to trial nurse by mobile telephone 9am - 5pm Monday-Friday for 12 weeks Trial nurse will - ensure FCP is appropriately shared with primary and secondary care, patient is registered on primary care palliative care register and will liaise with specialist PC services and the general practitioner as needed.

During the first 12 weeks of the study, patients randomised to usual care will not specifically receive these services. Recent audit from our centre suggests that delivery of such services to Heart Failure patients is inconsistent and generally poor while delivery of these services to people with coronary heart disease is non-existent.

Outcome-measures of the Phase 2 trial

Since this study is not powered to assess clinical outcomes, we plan to explore a number of outcomes that could be used in a later phase 3 trial. The following outcomes will be explored:

1. Patient and carer-centred outcomes:

   Outcomes will be assessed using the following questionnaire tools for both patients and their informer carers: ESAS - Edmonton symptom assessment scale, EQ5D - European Quality of Health Status, KDS - Kessler Distress Scale, Zarit 6 - caregiver burden questionnaire All patients will complete a series of questionnaires, addressing symptoms (Edmonton symptom assessment scale), quality of life (EQ5D) and distress (Kessler Distress scale) [20] immediately prior to discharge and at 6, 12, 18 and 24 weeks (see figure) and ideally within 7 days of each contact with the trial professionals. Since the intervention may have some impact on the carers we also plan to assess quality of life (EQ5D), distress (Kessler) and caregiver burden (Zarit 6) [21] using validated questionnaires at similar time points. Questionnaires will be mailed to the patient and carer approximately 2 days after each trial time point and the respondent will be encouraged to complete it within a further 3 days. The RA will offer telephone support to assist completion of these questionnaires in all cases to ensure consistency of response [22]. The RA will be responsible for the mailing, collection and collation of the outcome measures of the phase 2 trial and will be blinded to the randomisation status of the patient.
2. System outcomes All-cause unscheduled hospitalisation (including number of days in hospital), cardiovascular unscheduled hospitalisation, hospice admissions and use of other specialist palliative care services, achievement of primary care palliative care Quality Outcomes Framework criteria (placed on PC register, care plan in place and out of hours handover documented) by 6, 12 and 24 weeks after enrolment, whether the secondary and primary care case records contain documentation of care planning discussion and a formal record of CPR status at 6, 12, 18 and 24 weeks after enrolment. All patients will be followed up for 12 months after enrolment for hospitalisation outcomes.
3. After -death outcome measures These ill include assessment of time to death from study enrolment, cause of death, preferred place of care, actual place of death, Carer experience (VOICES questionnaire [22]). All patients will be followed up for 12 months following enrolment for mortality.

Data analysis and statistical issues Descriptive statistics (continuous variables: mean, standard deviation, median, range; categorical variables: number and percentage of participants) will be presented for the clinical and demographic features of the patients screened and those finally enrolled in the study. One of the main outcomes of our study which we will assess carefully is quality of life. The mean differences in EQ-5D health-related quality of life (QoL) utility between early and delayed intervention groups will firstly be analysed at the 12 week time point using analysis of covariance, adjusting for baseline utility score. We will then explore differences in QoL between groups at 24 weeks (t5) by the same method. The multiple measures at baseline, mid-point and end of intervention will allow analysis of trends in intervention effects on QoL and other parameters addressed by the distress and symptom assessment tools using repeated measures analysis of variance. The distribution and variability in EQ-5D values in this cohort of patients identified as having a poor prognosis will be used to inform the design and sample size of the future phase 3 trial. An economic evaluation in the phase 3 trial will consider, using a discrete choice experiment, patient preferences, values and willingness to pay for end of life care and the components which they value for quality of life. This approach complements the patient-centred nature of the intervention. Information to guide the design of the economic evaluation will be gathered using feedback from the qualitative component of this study.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years Unscheduled hospital admission due to congestive heart failure and or acute coronary syndrome 12 month estimated mortality risk of 20% or greater Optimal tolerated medical and device therapy

Exclusion Criteria:

Expected survival < 28 days Other life limiting non-cardiac condition likely to cause death within 12 months Moderate or severe dementia Moderate or severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6 months
  EuroQoL5D

SECONDARY OUTCOMES:
Hospital Readmissions | 6 months
  Unscheduled or non-elective admissions to hospital
Place of Death | 6 months
  Hospital, hospice or home
DNACPR status documented | 6 months
  Evidence of a discussion and agreed plan for Resuscitation Status of the patient
Mortality | 6 months
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Denvir, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Background] Denvir MA, Highet G, Robertson S, Cudmore S, Reid J, Ness A, Hogg K, Weir C, Murray S, Boyd K. Future Care Planning for patients approaching end-of-life with advanced heart disease: an interview study with patients, carers and healthcare professionals exploring the content, rationale and design of a randomised clinical trial. BMJ Open. 2014 Jul 14;4(7):e005021. doi: 10.1136/bmjopen-2014-005021. PMID 25023130
- [Derived] Anand A, Cudmore S, Robertson S, Stephen J, Haga K, Weir CJ, Murray SA, Boyd K, Gunn J, Iqbal J, MacLullich A, Shenkin SD, Fox KAA, Mills N, Denvir MA. Frailty assessment and risk prediction by GRACE score in older patients with acute myocardial infarction. BMC Geriatr. 2020 Mar 13;20(1):102. doi: 10.1186/s12877-020-1500-9. PMID 32164580